CLINICAL TRIAL: NCT05411549
Title: The Role of a Mediterranean Diet in Long-term Management of Pelvic Pain in Patients With Endometriosis: a Feasibility Trial
Brief Title: The Role of a Mediterranean Diet in Patients With Endometriosis: a Feasibility Trial
Acronym: MDIE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: McMaster - OBGYN - MDIE
Record Dates: First submitted 2022-03-28; First posted 2022-06-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis
Keywords: Diet Modification; Anti-Inflammatory Diet; Endometriosis Diet
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: 2 Arm Interventional Diet Modification Study Arm 1: Mediterranean Diet Counselling (Intervention) Arm 2: Continue Normal Diet (Control)
Who Masked: Participant, Outcomes Assessor
Masking Description: Data is de-identified upon collection, Lab teams will not be aware of arm allocation, nor will the participants be aware of the opposite group of which they are enrolled. However, due to the nature of this study, masking of the clinical team and participant is not feasible in order for diet changes to occur safely.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Experimental): Participants enrolled in group 1 will be counselled by a dietician and asked to adopt a Mediterranean diet for a 12-week period from counselling. Participants will complete the Mediterranean Diet Adherence Score, pain questionnaires as well as quality of life questionnaires (EPH-30, SF-36, GIQLI) which have been previously validated. Participants in this group will give a baseline and final visit blood sample and stool samples to assess inflammation biomarkers as well as gut microflora
  Interventions: Behavioral: Diet Modification to Adopt Mediterranean Diet
- No Diet Modification (No Intervention): Participants enrolled in group 2 will be NOT counselled by a dietician. Participants will complete the Mediterranean Diet Adherence Score, pain questionnaires as well as quality of life questionnaires (EPH-30, SF-36, GIQLI) which have been previously validated. Participants in this group will give a baseline and final visit blood sample and stool samples to assess inflammation biomarkers as well as gut microflora

INTERVENTIONS:
Behavioral: Diet Modification to Adopt Mediterranean Diet — Participants enrolled in group 1 will be counselled by a dietician and asked to adopt a Mediterranean diet for a 12-week period from counselling. Participants will complete a series of Mediterranean Diet Adherence Score, pain questionnaires as well as quality of life questionnaires (EPH-30, SF-36, GIQLI) which have been previously validated. Participants in this group will give a baseline and final visit blood sample and stool samples to assess inflammation biomarkers as well as gut microflora.
  Arms: Mediterranean Diet

SUMMARY:
This study aims to test if making changes to diet can affect the pelvic pain associated with endometriosis. One group will follow a Mediterranean diet for 12 weeks while the control group will continue with their current diet. We will be looking at the feasibility of a larger-scale trial as well as self-reported quality of life and self-reported pain using standardized questionnaires, that have previously been used and validated, and assessing how this diet affects biomarkers associated with endometriosis and inflammation. Further, we will test how this change in diet affects the gut microbe flora.

ELIGIBILITY:
Inclusion Criteria:

* Identified female at birth
* aged 18-45
* diagnosed with endometriosis (radiologically (ultrasound or magnetic resonance imaging (MRI)) or surgically confirmed diagnosis of endometriosis)
* Able and willing to provide written consent to participate in the study.

Exclusion Criteria:

* History of or diagnosis of gynecologic or GI malignancy
* Post-menopausal
* Currently pregnant or lactating
* Dietary restrictions due to medical conditions (e.g., Celiac disease, allergies)
* People who are already following a formal anti-inflammatory diet.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a large multi-site trial measured by assessing enrolment rate, dropout rate, time to sample size, adherence (Mediterranean Diet Adherence Score), time for intervention group to follow diet, food costs and frequency/type of Adverse Events. | 1 Year
  Dropout rate, time it takes to reach our sample size (24), adherence to the intervention using the Mediterranean Diet Adherence Score, the time it takes for study intervention group to be subjectively following the Mediterranean diet regularly, cost of food throughout the study, and frequency and type of Adverse Eventss will be measured using a case report form at each study visit.

SECONDARY OUTCOMES:
If the Mediterranean Diet improves pain of patients with endometriosis assessed using a visual analog scale (VAS) as well as the Endometriosis Health Profile (EHP-30). | 1 Year
  The VAS is measured on a 1 - 10 scale with 1 representing no pain and 10 representing life-debilitating pain.
  The EHP-30 is measured on a standardized scale from 0 to 100 where 0 represents the best health and 100 represents the worst health.
To assess whether the Mediterranean Diet can improve the concentration of peripheral inflammatory markers from baseline to study-end assessed using a 71 inflammatory marker protein array (EveTechnologies, Calgary, AB) | 1 Year
  Collection occurring at baseline and final visits
To assess if there is a change in the composition of the microbiota following a dietary change to the Mediterranean Diet using 16s ribosomal ribonucleic acid sequencing (McMaster Genomic Facility) | 1 Year
  Collection occurring at baseline and final visits

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Leonardi, M.D., Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No Identifiable information will be shared outside of the direct study team (clinical team, research coordinator). De-identification of all collected information will occur during collection as to not save personal identifiers in our database.